CLINICAL TRIAL: NCT04254185
Title: Clinical Trial for Surgery of the Ulnar Nerve (SUN) at the Elbow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Curtis National Hand Center (Unknown); Emory Healthcare (Other); Norton Healthcare (Other); Ohio State University (Other); OrthoCarolina Research Institute, Inc. (Other); University of Pittsburgh Medical Center (Other); Wake Forest University Health Sciences (Other); Johns Hopkins University (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Dr. Kevin C. Chung, Charles B de Nancrede Professor of Surgery, Professor of Surgery, Professor of Orthopaedic Surgery and Assistant Dean for Instructional Faculty, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00133613; U01AR073485 (NIH)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Neuropathy Ulnar
Keywords: Decompression; Anterior Subcutaneous Transposition; Elbow; Ulnar Nerve
MeSH Terms: conditions — Ulnar Neuropathies

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, multicenter, phase 3, randomized controlled superiority trial examining the treatment effectiveness of in-situ decompression and subcutaneous anterior transposition for UNE.
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simple decompression (Active Comparator): In-situ decompression releases only the compressive ligamentous structures overlying the ulnar nerve.
  Interventions: Procedure: Simple decompression
- Subcutaneous anterior transposition (Active Comparator): Anterior transposition repositions the ulnar nerve, providing decompression and lengthening by moving the nerve anterior to the axis of elbow rotation
  Interventions: Procedure: Subcutaneous anterior transposition

INTERVENTIONS:
Procedure: Simple decompression — Surgical technique
  Other Names: In-situ Decompression
  Arms: Simple decompression
Procedure: Subcutaneous anterior transposition — Surgical technique
  Arms: Subcutaneous anterior transposition

SUMMARY:
This research is studying two surgical procedures in a large group of people to learn about how well these procedures work as a treatment for ulnar neuropathy at the elbow (UNE). Researchers want to see which surgery is more helpful for people with ulnar neuropathy. This research will determine if one surgery is better than the other to alleviate symptoms.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis or suspected diagnosis of isolated ulnar neuropathy at the elbow
* Confirmation of ulnar neuropathy using the American Association of Electrodiagnostic Medicine criteria for electrodiagnostic studies at the elbow. (Participants must meet at least 1 of the criteria to be enrolled (absolute motor nerve conduction from above elbow (AE) to below elbow (BE) of less than 50 m/s; An AE to BE segment greater than 10 m/s slower than BE to wrist segment; A decrease in compound muscle action potential (CMAP) negative peak amplitude from BE to AE greater than 20%)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Able to read, understand and complete the questionnaires in English

Exclusion Criteria:

* Previous elbow fracture requiring surgical fixation
* Patients who have not attempted conservative management for UNE (e.g. night splinting)
* Subluxation of ulnar nerve on preoperative exam
* Recurrent UNE after previous surgery
* Concomitant neuropathic conditions such as Carpal Tunnel Syndrome or cervical or brachial plexus abnormalities
* Participants with severe comorbid conditions that prohibit surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of surgery as measured by the Michigan Hand Outcomes Questionnaire (MHQ) summary score | 1 year
  The MHQ is a self-report measure that assesses the function of the hand(s) and/or wrist(s). The MHQ contains six distinct scales assessing overall hand function, activities of daily living, pain, work performance, aesthetics and subject satisfaction with hand function. Scores range from 0-100, 100=no disability). In the pain scale, however, high scores indicate greater pain (0-100, 0=no pain).

SECONDARY OUTCOMES:
Recovery as measured by the Michigan Hand Outcomes Questionnaire (MHQ) pain score | Up to 1 year
  The MHQ is a self-report measure that assesses the function of hand(s) and/or wrist(s). The MHQ contains six distinct scales. The score will be measured at various time points to identify the recovery trend.In a pain scale, high scores indicate greater pain (0-100, 0=no pain)
Recovery as assessed by the Carpal tunnel questionnaire (CTQ) symptom score | Up to 1 year
  The CTQ (also known as the Levine Questionnaire, Boston Questionnaire, and the Brigham and Women's Questionnaire) contains 19 questions (11 symptom severity questions and 8 functional status questions). All questions use a scale of 1 to 5, with 1 being the best score or no symptoms.
  The score will be measured at various time points to identify the recovery trend.
Recovery as assessed by the Carpal tunnel questionnaire (CTQ) pain score | Up to 1 year
  The CTQ (also known as the Levine Questionnaire, Boston Questionnaire, and the Brigham and Women's Questionnaire) contains 19 questions (11 symptom severity questions and 8 functional status questions). All questions use a scale of 1 to 5, with 1 being the best score or no symptoms.
  The score will be measured at various time points to identify the recovery trend.
Difference in Grip Strength (unaffected hand - affected hand) measured by a Jamar dynamometer | Up to 1 year
  Measured in kilograms. Grip strength will be measured at various time points to identify the recovery trend.
Difference in Pinch Strength (unaffected hand - affected hand) as measured by a pinch gauge | Up to 1 year
  Pinch strength will be recorded, to the nearest half-kilogram. It will be measured at various time points to identify the recovery trend.
Difference in distance assessed by the 2 Point Discrimination (unaffected hand - affected hand) | Up to 1 year
  Thresholds on the tip of the finger of both hands are assessed using the method of constant stimuli. One single needle and seven pairs of needles with different spacing's are tested in randomized order. After each presentation, the subject has to report the sensation of one or two needles by answering immediately "one" or "two." The threshold difference will be measured at various time points to identify the recovery trend.
Sensory difference as assessed by Semmes-Weinstein Monofilament test (unaffected hand - affected hand) | Up to 1 year
  A quantitative method to systematically assess the threshold stimulus necessary for perception of light touch to deep pressure by using monofilaments of different sizes.
  Interpretation scale for monofilaments:
  2.83 Normal 3.61 Diminished light touch 4.31 Diminished protective sensation 4.56 Loss of protective sensation 6.65 Deep pressure sensation only Sensory thresholds will be measured at various time points to identify the recovery trend.
Complication rates for both surgical procedures assessed using a checklist | Up to 1 year
  Complications will be categorized by type, severity, and frequency captured at Surgery, 2-Week, 6-Week, 3-Month, and 12 Month Visits.
Disease severity as measured by ulnar neuropathy at the elbow (UNE) severity scale | Enrollment, approximately day 0
  Severity is determined based on responses to three parts sensory, motor, and test outcomes. Each part is scored 1-3, where 3=most disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Chung, MD, MS, Principal Investigator — University of Michigan
Locations (10):
- United States (10):
  - Emory Healthcare, Atlanta, Georgia
  - Norton Healthcare, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Curtis National Hand Center, Baltimore, Maryland
  - Michigan Medicine, Ann Arbor, Michigan
  - OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung KC, Malay S, Burns PB, Kim HM, Ki J; SUN Study Group. Predictors of disease severity for ulnar neuropathy at the elbow, analysis from a randomized clinical trial. Plast Reconstr Surg. 2025 Sep 23. doi: 10.1097/PRS.0000000000012472. Online ahead of print. PMID 40991254